CLINICAL TRIAL: NCT07083778
Title: A Randomized Controlled Trial to Determine the Efficacy and Safety of Laser Versus Open Surgery in the Treatment of Fistula-in-Ano at a Tertiary Care Centre
Brief Title: Comparison Between Laser and Open Fistula Surgeries in the Management of Fistula - In - Ano
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GSVM Medical College (Other)
Responsible Party: Principal Investigator, Kamal raj, Junior Resident , Department of general Surgery, GSVM Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GSVM-FIA-RCT-2025-01
Record Dates: First submitted 2025-07-02; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: FISTULA IN ANO
Keywords: Fistula-in-ano; Laser fistula surgery; Fistulotomy; Fistulectomy; Postoperative pain; Healing rate; Randomized controlled trial; Recurrence; Incontinence; Intersphincteric fistula; Transsphincteric fistula
MeSH Terms: conditions — Rectal Fistula; Pain, Postoperative; Recurrence

STUDY DESIGN:
Intervention Model Description: This study is a prospective, single-center, randomized controlled trial designed to compare the efficacy and safety of laser ablation (FiLaC technique) versus conventional open surgical techniques (fistulotomy/fistulectomy) in patients diagnosed with intersphincteric or transsphincteric fistula-in-ano.
  Patients were randomly assigned in a 1:1 ratio to undergo either laser surgery or open surgery after evaluation through clinical examination and MR fistulogram. Both groups were managed as per standard operative protocols and followed up for a period of three months.
  The study assessed both clinical outcomes and patient-reported outcomes, including postoperative pain (VAS score), duration of hospital stay, time to resume daily activities, healing rate, recurrence, postoperative complications (like incontinence, wound infection), and overall patient satisfaction.
  This model evaluates the utility of a minimally invasive sphincter-preserving laser technique in comparison to the tradition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental - Laser Surgery Group (Experimental): Patients randomized to this arm will undergo laser ablation of the fistula tract using a radial fiber laser probe (e.g., FiLaC technique). The procedure is performed under spinal or general anesthesia. The internal opening is closed, and laser energy (10W in pulsed mode) is delivered circumferentially along the fistula tract to ablate it.
  All patients will receive standard perioperative care, including IV antibiotics preoperatively and oral antibiotics postoperatively.
  Interventions: Procedure: Laser Fistula Surgery (FiLaC - Fistula-tract Laser Closure)
- Active Comparator - Open Surgery Group (Active Comparator): Patients randomized to this arm will undergo standard open surgery (fistulotomy or fistulectomy or LIFT ), depending on the anatomy of the fistula. The tract will be laid open or excised under spinal anesthesia. Wounds will be left to heal by secondary intention.
  Standard postoperative care includes oral antibiotics, analgesia, sitz baths, and regular dressings.
  Interventions: Procedure: Open Fistula Surgery (Fistulotomy, Fistulectomy, or LIFT Procedure)

INTERVENTIONS:
Procedure: Laser Fistula Surgery (FiLaC - Fistula-tract Laser Closure) — A minimally invasive procedure using a radial fiber diode laser probe to ablate the fistula tract. Laser energy (10W in pulsed mode) is applied circumferentially as the probe is slowly withdrawn, leading to shrinkage and closure of the fistula tract. The internal opening is closed with absorbable sutures. The procedure is done under spinal or general anesthesia.
  Arms: Experimental - Laser Surgery Group
Procedure: Open Fistula Surgery (Fistulotomy, Fistulectomy, or LIFT Procedure) — Patients in this group will undergo standard open surgical treatment for fistula-in-ano. Based on the type and location of the fistula (intersphincteric or transsphincteric), the surgical procedure may be:
  * Fistulotomy: Laying open the fistula tract.
  * Fistulectomy: Excision of the entire fistulous tract.
  * LIFT Procedure: Ligation of the intersphincteric fistula tract, preserving the sphincter complex. This sphincter-sparing technique is chosen for transsphincteric fistulas when appropriate.
  All procedures are performed under spinal anesthesia. The choice of technique is individualized based on MR fistulogram findings and intraoperative assessment. Wounds are managed with regular dressings and allowed to heal by secondary intention. Standard postoperative care includes antibiotics, analgesia, and sitz baths. Follow-up is done at 1 week, 1 month, 3 months, and 6 months.
  Arms: Active Comparator - Open Surgery Group

SUMMARY:
This prospective randomized controlled trial compared the outcomes of laser versus open surgical techniques in the management of fistula-in-ano among 100 patients at a tertiary care center. Patients were diagnosed with intersphincteric or transsphincteric fistulas using clinical examination and MR fistulogram and were randomly assigned to undergo either laser surgery (n=50) or open surgery (n=50).

The primary endpoints included postoperative pain, hospital stay duration, and time to return to normal activity. Secondary outcomes assessed were recurrence, wound infection, incontinence, need for reoperation, and patient satisfaction.

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label, parallel-group interventional clinical trial conducted at GSVM Medical College, Kanpur, aimed at comparing the clinical efficacy and safety of laser surgery using the FiLaC (Fistula Laser Closure) technique versus conventional open surgical procedures (fistulotomy or fistulectomy) in the management of fistula-in-ano.

A total of 100 adult patients (>18 years), with a confirmed diagnosis of intersphincteric or transsphincteric fistula-in-ano based on clinical evaluation and magnetic resonance (MR) fistulogram, were enrolled. Following informed consent and screening, patients were randomized in a 1:1 ratio into two arms:

Group A (Laser Surgery Group): Underwent minimally invasive FiLaC procedure using a 1470 nm diode laser and radial fiber probe for endofistular ablation.

Group B (Open Surgery Group): Underwent traditional open surgical procedures including fistulotomy, fistulectomy, or LIFT (Ligation of Intersphincteric Fistula Tract), depending on fistula anatomy.

All surgeries were performed under spinal anesthesia. Postoperative care was standardized across both groups. Patients were followed for a minimum of 3 months with structured clinical assessments at regular intervals.

Primary outcome measures included:

Postoperative pain (VAS score within 7 days)

Duration of hospital stay

Time to resume normal daily activity

Secondary outcomes evaluated were:

Recurrence rate at 3 months

Complete healing within 3 months (closure of both internal and external openings, cessation of discharge)

Anal incontinence rate

Anal stenosis rate

The study intends to assess whether the laser approach offers a meaningful improvement in postoperative morbidity, patient comfort, and quality of life, while also examining risk factors associated with poor surgical outcomes or recurrence.

ELIGIBILITY:
Inclusion Criteria:

* • Patient with intersphincter & transphincter fistula in ano as confirmed by clinical examination followed by MR fistulogram.

  * Age 18 to 65 years
  * Non responders and Recurrent Patient giving written informed consent of selected fistula surgery and having awareness about alternative procedures.

Exclusion Criteria:

* • Pregnant women

  * Patients of fistula in ano associated with other conditions(HIV, tubercular disease, IBD, Ca rectum.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain at 48 Hours | 48 hours post-surgery
  Assessment of postoperative pain using the Visual Analogue Scale (VAS) scored from 0 (no pain) to 10 (worst pain imaginable), recorded at 48 hours after surgery.
Length of Hospital Stay | From day of surgery to discharge (typically within 7 days)
  Total number of days the patient remains admitted in the hospital from the day of surgery until discharge.
Time to Return to Normal Work | Within 6 weeks post-surgery
  Number of days taken by the patient to resume normal daily activities or work, as self-reported during follow-up visits.

SECONDARY OUTCOMES:
Fistula Recurrence Rate | Between 16 to 20 weeks post-surgery
  Proportion of patients showing recurrence of fistula-in-ano after surgery, confirmed clinically or radiologically.
Time to Complete Healing | Within 3 months post-surgery
  Number of days from surgery to complete wound healing, defined as epithelialization of the surgical site without discharge.
Anal Incontinence Rate (Wexner Score) | Assessed at each follow-up up to 6 months
  Incidence of anal incontinence assessed using the Wexner Incontinence Score, a validated scale ranging from 0 (perfect continence) to 20 (complete incontinence).
Anal Stenosis Rate | Within 3 months post-surgery
  Proportion of patients developing clinically significant anal stenosis, defined as narrowing of the anal canal requiring intervention or causing obstructive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Raj, MS surgery, Principal Investigator — GSVM MEDICAL COLLEGE , KANPUR
Locations (1):
- Kamal Raj, Kanpur, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual-level data related to primary and secondary outcomes.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication of the main results, for up to 5 years.
Access Criteria: Qualified researchers upon reasonable request.
URL: http://gsvmmedicalcollege.com

REFERENCES:
- [Derived] Patel KR, Jauhari RK, Shukla P. A Randomized Controlled Trial Comparing Laser Versus Open Surgical Approaches in the Management of Fistula-in-Ano at a Tertiary Care Center. Cureus. 2025 Aug 19;17(8):e90471. doi: 10.7759/cureus.90471. eCollection 2025 Aug. PMID 40978994

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT07083778/Prot_SAP_000.pdf